CLINICAL TRIAL: NCT02785276
Title: Intra-abdominal Infusions of Ropivacaine Following Laparoscopic Ventral Hernia Repair: a Randomised Double-blind Controlled Trial.
Brief Title: Improving Pain Relief Following Laparoscopic Ventral Hernia Repair
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study not initiated
Sponsor: University of Auckland, New Zealand (Other)
Responsible Party: Principal Investigator, Andrew G Hill, MBChB, MD (Thesis), EdD, FACS, FRACS, Professor of Surgery, University of Auckland, New Zealand
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: COLVHR
Record Dates: First submitted 2016-05-23; First posted 2016-05-27 (Estimated); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Pain, Postoperative; Anesthesia, Local; Hernia, Ventral; Laparoscopy; Analgesics, Opioid; Complications
MeSH Terms: conditions — Pain, Postoperative; Hernia, Ventral | interventions — Ropivacaine; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ropivacaine infusion (Experimental): Following the insertion of the 2mm fenestrated catheter, the wound catheter will be connected to the 270mL AutoFuser Pain Pump. The intraperitoneal infusion with ropivacaine (0.2%) at 4 mL/hour will start immediately and continue for 68 hours post-operatively uninterrupted.
  Interventions: Device: AutoFuser Pain Pump; Drug: Ropivacaine
- Placebo infusion (Placebo Comparator): In the same manner as described for the ropivacaine infusion arm, 0.9% Normal Saline will be administered over 68 hours.
  Interventions: Device: AutoFuser Pain Pump; Other: Normal Saline (0.9%)

INTERVENTIONS:
Device: AutoFuser Pain Pump — Closed loop local anaesthetic infusion system
Drug: Ropivacaine — Commonly used local anaesthetic drug
  Other Names: Naropin (0.2%)
  Arms: Ropivacaine infusion
Other: Normal Saline (0.9%) — Normal saline is a sterile, non-pyrogenic solution for fluid and electrolyte replenishment for intravenous administration. This will be the solution used for the intraperitoneal infusion in the placebo/control group.
  Other Names: Sodium chloride (NaCl)
  Arms: Placebo infusion

SUMMARY:
Aim

The general aim of this study is to improve post-operative pain and reduce morphine consumption following laparoscopic ventral hernia repair (LVHR). We specifically aim to conduct a randomized, double blinded, controlled trial to investigate the effect of intra-peritoneal local anaesthesia infusions on post-operative morphine consumption and.

Methods:

Patients will be randomised by computer generated random numbers (random permutation) and opaque envelope methods. At closure, one small 2mm catheter belonging to the AutoFuser pain pump system will be placed in the peritoneal cavity between the onlay mesh and parietal peritoneum. In the treatment arm patients will receive 275mL of 0.2% ropivacaine at 4mL/h. In the placebo arm, 275mL of 0.9% normal saline will be used in a similar fashion. The infusions will run for 68 hours total. All members involved in patient care (with the exception of one independant research fellow) will be blinded to the above. After 68 hours the pump will be stopped and the catheter will be removed. Assessment of post-operative pain will be performed by visual analogue scale, and total opiate consumption will be collected and converted into morphine equivalents.

Health significance:

Local anaesthesia has become an important addition to multimodal regimens of analgesia following surgery. Recent studies have shown that local anaesthetic (LA) wound infiltration has improved post-operative pain when compared with standard opioid regimens for pain relief. Only one previous study looked at bupivacaine infusions into the hernia sac for three days following LVHR. This study found no improvement in post-operative pain or morphine consumption. We aim to demonstrate improved pain and reduced morphine consumption using an alternative catheter insertion technique and ropivacaine as the desired LA agent.

DETAILED DESCRIPTION:
Scientific background:

A ventral hernia (VH) is a fascial defect located in the anterior abdominal wall. Primary VH includes epigastric, umbilical and spigelian hernias. A secondary defect or incisional hernia develops at a previous surgical incision site (1). VHs are a common condition and risk factors include obesity, previous abdominal surgery and elevated intra-abdominal pressure (2). With New Zealand's rising obesity epidemic the incidence of VH is projected to increase (3-4). Optimising the peri-operative care of patients undergoing VH repair is critical to cost-effective healthcare of this increasingly significant issue.

Surgical repair aims to relieve symptoms and prevent complications (5-6). Open mesh repair has been the accepted gold standard since proving superior to open suture repair (7). Laparoscopic ventral hernia repair (LVHR) has grown in popularity since its introduction in 1993 (8). Studies have shown advantages over open repair such as fewer infectious complications and shorter hospital stay (9-12). Importantly, LVHR is favourable in obese patients (BMI>30) due to lower complication rates and overall cost of care (13-16). Laparoscopic surgery has been considered less painful in comparison to open surgery, yet trials report no difference in acute or chronic pain (17-19). Severe pain following LVHR is a significant clinical problem impacting on wellbeing, quality of life and patient satisfaction (20). One hypothesis to explain this pain is the use of tacks and sutures for mesh fixation (21-23).

Local anaesthesia has become a key adjunct to multimodal post-operative regimens of analgesia. This is due to fewer side effects such as nausea and vomiting, gut dysmotility and respiratory depression (24). Local anaesthetic (LA) agents are easily applied directly to the injury site blocking afferent nociceptive nerves and reducing the local inflammatory response (25). There are significant benefits to intraperitoneal application of LA agents following abdominal surgery (26-27). Hence, operative insult to the peritoneum following LVHR may be controlled with LA directed to the site of mesh fixation in the intraperitoneal cavity (28).

Objective:

Conduct a randomised double-blinded controlled trial to investigate the effect of intra-peritoneal local anaesthesia infusions on post-operative pain and morphine consumption in patients undergoing LVHR.

Research Design:

Randomised double-blinded clinical trial to investigating intra-peritoneal infusions of ropivacaine on post-operative pain scores in patients undergoing LVHR procedures.

Ethics:

Ethics approval for this project is yet to be obtained.

Sample size:

Using morphine consumption data from a retrospective study we conducted in evaluating the total opiate consumption in the first 24 hours following LVHR surgery, in order to detect a reduction of morphine consumption by 50% in the first 24 hours post-operatively with alpha of 0.05 and power of 0.9, 43 patients are required in each group. We will aim for 48 patients in each arm anticipating for possible drop outs.

Methodology:

Patients will be recruited from surgical outpatient clinics at Manukau Super Clinic (MSC). Patients who are undergoing LVHR will be invited to partake in the study. As the research fellow in this study I will be involved in data collection and data analysis.

Patients will be randomised by computer generated random numbers and opaque envelope methods. In the treatment arm patients will receive 275mL of 0.2% ropivacaine after wound catheter insertion or in the placebo arm, receive 275mL of 0.9% normal saline in a similar fashion. One theatre staff nurse who will not be involved in patient care will be given the blinded envelope and the pre-prepared lidocaine or saline mixtures in the theatre drug room. The mixtures will be unlabelled and appear similar in color. All members of the staff involved in patient care including the anaesthetist will be blinded to the solution administered. The theatre staff nurse will then prepare a small infusion pump (AutoFuser). The mixture used in the pump will be pre-mixed by one of the clinical pharmacists at Middlemore hospital who will not be involved in patient care. The staff nurse will be un-blinded to the contents of the mixtures. The nurse will prepare the pump and load either the local anaesthetic or saline solution. At closure, one small 2mm catheter, with 30 small fenestrations at the end, will be placed in the peritoneal cavity between the onlay mesh and parietal peritoneum to infuse local anaesthetic. This will penetrate through the skin once closure is complete. This will be attached to the infusion pump (AutoFuser). This pump will contain either 270mls of 0.2% ropivacaine or 270mls of 0.9% saline. All members involved in patient care including surgical, anaesthetic and nursing teams will be blinded to the contents of this pump. The pump will be activated at a set rate of 4mls/hr immediately once the patient is in the post-anaesthesia recovery room. The pump will run continuously. The patient will continue recovery on the ward as per the surgical team. After 68 hrs the pump will be stopped and the catheter will be removed in a similar fashion as routine drain removal.

Endpoints:

1. Assessment of post-operative pain using Visual analogue scale (VAS) 1 hour, 2 hours, 4 hours, 6 hours, 8 hours, day 1, day 2 and day 3 post operatively.
2. Total opiate consumption in the first 24 hours (manually converted to morphine equivalents)

Resources:

Consultant General Surgeons at Middlemore Hospital

Consultant anaesthetist: Dr. Nicholas Lightfoot

Patients: approximately 85 LVHR procedures are performed at MSC per year.

Manukau Surgical Centre staff facilities

University of Auckland facilities

AutoFuser pain pumps

Ropivacaine (0.2%) - Naropin

Normal Saline (0.9)

ELIGIBILITY:
Inclusion Criteria:

* All consecutive consenting adult patients (≥16 years) undergoing elective LVHR (umbilical / incisional / spigelian) will be screened for inclusion

Exclusion Criteria:

* acute presentation, open repair of ventral hernia, hepatic dysfunction ALT/AST ≥ 2 x ULN, previous adverse reaction/allergy to ropivacaine, opiate use greater than 6 months, patients with a diagnosis of Chronic Pain Syndrome (CPS), patients under 16 years of age, patient refusal and those without the ability to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-08; Primary Completion 2017-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Morphine equivalent use | Total opiate consumption in the first 24 hours
  Total opiate analgesia (all routes) used from immediately post-operative (0h) during the post-operative recovery period up to 24 hours will be recorded and converted into morphine equivalents.

SECONDARY OUTCOMES:
Post-operative pain scores | Until day 7 post-operatively
  Abdominal pain at rest, on moving (recumbent to the upright position), and on coughing will be assessed using 3 separate 10 point Visual Analogue Scales (VAS) preoperatively (baseline), at 2, 4, 6, 8, 12, 24, 48 and 72 hours as well as on day 7 postoperatively

OTHER OUTCOMES:
Complications | From immediately post-operative up until 30 days following laparoscopic ventral hernia repair
  Postoperative 30 day-complication rates will be recorded prospectively. All complications (including multiple occurrences per patient) will be recorded, pooled and graded as per the Clavien- Dindo classification system

CONTACTS AND LOCATIONS:
Overall Officials: Andrew G Hill, MD, EdD, FACS, FRACS, Principal Investigator — The University of Auckland
Locations (1):
- Manukau Surgical Centre, Middlemore Hospital, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No